CLINICAL TRIAL: NCT01789320
Title: Open-Label, Safety and Tolerability Study of Suprachoroidal Triamcinolone Acetonide Via Microneedle in Subjects With Non-Infectious Uveitis
Brief Title: Safety Study of Suprachoroidal Triamcinolone Acetonide Via Microneedle to Treat Uveitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Clearside Biomedical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLS1001-101
Record Dates: First submitted 2013-02-05; First posted 2013-02-12 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Uveitis; Intermediate Uveitis; Posterior Uveitis; Panuveitis; Noninfectious Uveitis
Keywords: uveitis; intermediate uveitis; posterior uveitis; panuveitis; noninfectious uveitis; microneedle; suprachoroidal space; SCS; inflammation; ocular inflammatory conditions; triamcinolone acetonide; TA; Triesence; injection; IVT; intravitreal; corticosteroid; sympathetic ophthalmia; temporal arteritis; vitreous haze
MeSH Terms: conditions — Uveitis; Uveitis, Intermediate; Uveitis, Posterior; Panuveitis; Choroidal Effusions; Inflammation; Ophthalmia, Sympathetic; Giant Cell Arteritis | interventions — Triamcinolone Acetonide; Triamcinolone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- triamcinolone acetonide (Triesence®) (Experimental): TRIESENCE® (triamcinolone acetonide injectable suspension 40 mg/mL) in a total volume of 100 uL administered via microneedle directly to the suprachoroidal space (SCS)
  Interventions: Drug: triamcinolone acetonide (Triesence®)

INTERVENTIONS:
Drug: triamcinolone acetonide (Triesence®) — 4 mg of TRIESENCE® (triamcinolone acetonide injectable suspension 40 mg/mL) administered as a single injection to the suprachoroidal space
  Other Names: triamcinolone acetonide; TA; Triesence; corticosteroid

SUMMARY:
This study is designed to determine the safety and tolerability of a single microinjection of triamcinolone acetonide (TRIESENCE®) into the suprachoroidal space (SCS) of patients who have non-infectious uveitis.

DETAILED DESCRIPTION:
This is a Phase 1/2, open-label study designed to evaluate the safety, tolerability and procedure of a microneedle injection of triamcinolone acetonide (TA) into the SCS. The subjects enrolled in this study will be chosen from subjects with non-infectious intermediate, posterior and pan-uveitis. The injection will only be administered to a single eye via the Clearside Biomedical proprietary microneedle into the SCS. The dose of TA to be injected is 4 mg of currently approved TRIESENCE® (triamcinolone acetonide injectable suspension 40 mg/mL). The study design includes 10 clinic visits over 27 weeks. Subjects will be followed for 26 weeks following treatment with TRIESENCE®.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of non-infectious intermediate, posterior or pan-uveitis

Exclusion Criteria:

* any ocular trauma within the past 6 months in the study eye
* any injection of intraocular corticosteroids or steroid implant or the Ozurdex® implant in the 6 months prior to the study treatment, or any prior use of Retisert™ in the study eye
* any uncontrolled systemic disease that would preclude participation in the study or put the subject at risk due to study treatment or procedures
* have a known HIV infection or other immunodeficiency disease for which corticosteroid therapy would be contraindicated
* are monocular
* have ocular hypertension
* history of any intraocular surgery in the study eye
* presence of an anterior staphyloma in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Ciulla, MD, Study Director — Clearside Biomedical, Inc.
Locations (3):
- United States (3):
  - Northwestern University, Chicago, Illinois
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Cleveland Clinic Foundation, Cleveland, Ohio

REFERENCES:
- [Derived] Goldstein DA, Do D, Noronha G, Kissner JM, Srivastava SK, Nguyen QD. Suprachoroidal Corticosteroid Administration: A Novel Route for Local Treatment of Noninfectious Uveitis. Transl Vis Sci Technol. 2016 Dec 14;5(6):14. doi: 10.1167/tvst.5.6.14. eCollection 2016 Dec. PMID 27980877

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Triamcinolone Acetonide (Triesence®)
Started | 11
Completed | 9
Not Completed | 2
Not completed — Re-enrolled into study | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All subjects who received at least one attempted dose of study drug.
Arm/Group | Triamcinolone Acetonide (Triesence®)
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (9.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 4
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure (IOP)
Description: Intraocular pressure is the fluid pressure inside the eye. Intraocular pressure change from baseline at week 8 was measured by Goldmann applanation tonometry. Tonometry is the method eye care professionals use to determine this pressure. Intraocular pressure is typically measured in millimeters of mercury. A higher pressure inside the eye can be a risk factor for developing glaucoma or glaucoma progression leading to optic nerve damage. A negative change indicates a reduction in intraocular pressure.
Time Frame: Change from baseline in IOP at 8 weeks
Population: Safety population including all subjects who received at least one attempted dose of study drug.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Triamcinolone Acetonide (Triesence®)
Number analyzed (Participants) | 10
mm Hg | -0.1 (3.21)

2. Primary Outcome: Best Corrected Visual Acuity
Description: Visual acuity (VA) rates a person's ability to recognize small details with precision. Best corrected VA refers to this measurement when the best vision has be achieved following refraction. Visual acuity change from baseline at 8 and 26 weeks was measured following the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol using standardized lighting and lanes and an ETDRS eye chart. This eye chart comprises rows of letters, with 5 letters per row, and with the letter size from line to line varying logarithmically and is used to estimate visual acuity. Visual acuity is scored with reference to the logarithm of the minimum angle of resolution or logMAR. Zero logMAR indicates standard vision, positive values indicate poor vision and negative values indicate good vision. A negative changes indicates an improvement in visual acuity.
Time Frame: Change from baseline at 8 weeks and 26 weeks.
Population: Per protocol population including all subjects who received at least one attempted dose of study drug. Data post-rescue was excluded.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Triamcinolone Acetonide (Triesence®)
Number analyzed (Participants) | 8
logMAR
  Week 8 | -0.25 (0.107)
  Week 26: number analyzed (Participants) | 4
  Week 26 | -0.28 (0.096)

3. Secondary Outcome: Central Subfield Thickness Using Optical Coherence Tomography (OCT)
Description: Central subfield thickness (CST) is a measure of the thickness of the retina in the 1 mm diameter circle centered on the fovea or center of the macular where eyesight is the sharpest. CST change from baseline at 8 and 26 weeks was measured using optical coherence tomography (OCT). OCT is a diagnostic imaging technique used to capture 2 and 3 dimensional images within biological tissue, e.g., for determining the amount of edema contained in the retina. CST is typically measured in microns. A negative change represents a reduction in retinal thickness and an improvement in cases of retinal edema.
Time Frame: Change from baseline at 8 weeks and 26 weeks.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Triamcinolone Acetonide (Triesence®)
Number analyzed (Participants) | 7
Microns
  Week 8 | -153.7 (109.45)
  Week 26: number analyzed (Participants) | 3
  Week 26 | -107.0 (86.95)

4. Secondary Outcome: Vitreous Haze Grade
Description: Vitreous haze scale (Nussenblatt 1985 as modified in Lowder 2011). Scores include value 0 (no inflammation), +0.5 (trace inflammation), +1 (mild blurring of the retinal vessels and optic nerve), +1.5 (optic nerve head and posterior retina view obscuration greater than +1 but less than +2), +2 (moderate blurring of the optic nerve head), +3 (marked blurring of the optic nerve head), and +4 (optic nerve head not visible) A higher score indicates a worse outcome.
Time Frame: Change from baseline at 8 weeks and 26 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triamcinolone Acetonide (Triesence®)
Number analyzed (Participants) | 8
score on a scale
  Week 8 | -0.75 (0.463)
  Week 26: number analyzed (Participants) | 4
  Week 26 | -0.75 (0.289)

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Triamcinolone Acetonide (Triesence®)
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triamcinolone Acetonide (Triesence®) (N=11)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triamcinolone Acetonide (Triesence®) (N=11)
Cataract (Eye disorders) | 1 (1) — #Study eye
Cystoid macular oedema (Eye disorders) | 3 (3) — #Study eye
Cystoid macular oedema (Eye disorders) | 1 (1) — #Fellow eye
Eye irritation (Eye disorders) | 1 (1) — #Study eye
Eye pain (Eye disorders) | 5 (6) — #Study eye
Eyelid margin crusting (Eye disorders) | 1 (1) — #Study eye
Punctate keratitis (Eye disorders) | 1 (1) — #Study eye
Retinal ischaemia (Eye disorders) | 1 (1) — #Study eye
Retinal neovascularisation (Eye disorders) | 1 (1) — #Study eye
Uveitis (Eye disorders) | 1 (1) — #Study eye
Vision blurred (Eye disorders) | 1 (2) — #Study eye; both events occurred in a subject who received 0 µL of study drug.
Visual acuity reduced (Eye disorders) | 2 (2) — #Study eye
Visual acuity reduced (Eye disorders) | 1 (1) — #Fellow eye
Pyrexia (General disorders) | 1 (1) — #Event occurred in a subject who received 0 µL of study drug.
Localised infection (Infections and infestations) | 2 (2) — #Both events occurred in a subject who received 0 µL of study drug.
Sinusitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) — #Event occurred in a subject who received 0 µL of study drug.
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) — #Event occurred in a subject who received 0 µL of study drug.
Headache (Nervous system disorders) | 2 (3)
Psychological trauma (Psychiatric disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) — #Event occurred in a subject who received 0 µL of study drug.
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Cataract operation (Surgical and medical procedures) | 1 (1) — #Study eye; event occurred in a subject who received 0 µL of study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The institution and investigators participating in this trial shall have no right to publish or present the results of this study without the prior written consent of Clearside Biomedical (or designee).